CLINICAL TRIAL: NCT02648438
Title: An Open Label, Partially Randomized, Four-period Study in Healthy Male Subjects to Investigate the Bioavailability and Pharmacokinetics of a Single Dose of AZD7594 When Administered Intravenously, Orally and Inhaled Via Two Different Dry Powder Inhalers (DPI) and a Pressurized Metered-dose Inhaler (pMDI)
Brief Title: A Study to Assess the Bioavailability and to Compare the Pharmacokinetics of AZD7594 Inhaled Via Monodose Inhaler and Multiple-dose Dry Powder Inhalers (DPI) or Pressurized Metered-dose Inhaler (pMDI) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D3741C00004
Record Dates: First submitted 2015-12-26; First posted 2016-01-07 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-03

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: AZD7594; Bioavailability; Healthy male subjects; Safety; Tolerability; Pharmacokinetics; Monodose inhaler; Multiple-dose dry powder inhaler
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence 1 (Experimental): Treatment Period 1:AZD7594 Solution for infusion (150 μg intravenous formulation) Treatment Period 2:AZD7594 Inhalation powder (400 μg) by dry powder inhaler (DPI) Device 1 (monodose inhaler) Treatment Period 3:AZD7594 Inhalation powder (400 μg) by DPI device 2 (multiple-dose inhaler) Treatment Period 4:AZD7594 Oral suspension (1200 μg oral formulation)
  Interventions: Drug: AZD7594 Solution for infusion (150 μg intravenous formulation); Drug: AZD7594 Oral suspension (1200 μg oral formulation); Drug: AZD7594 Inhalation powder (400 μg) by DPI Device 1 (monodose inhaler); Drug: AZD7594 Inhalation powder (400 μg) by DPI device 2 (multiple-dose inhaler)
- Treatment sequence 2 (Experimental): Treatment Period 1:AZD7594 Solution for infusion (150 μg intravenous formulation) Treatment Period 2:AZD7594 Inhalation powder (400 μg) by dry powder inhaler (DPI) Device 1 (monodose inhaler) Treatment Period 3:AZD7594 Pressurized inhalation suspension (400 μg) by pressurized metered-dose inhaler (pMDI) Treatment Period 4:AZD7594 Oral suspension (1200 μg oral formulation)
  Interventions: Drug: AZD7594 Solution for infusion (150 μg intravenous formulation); Drug: AZD7594 Oral suspension (1200 μg oral formulation); Drug: AZD7594 Inhalation powder (400 μg) by DPI Device 1 (monodose inhaler); Drug: AZD7594 Pressurized inhalation suspension (400 μg) by pMDI

INTERVENTIONS:
Drug: AZD7594 Solution for infusion (150 μg intravenous formulation) — Solution for infusion 0.01 mg/ml; AZD7594 150 μg IV
Drug: AZD7594 Oral suspension (1200 μg oral formulation) — 0.1 - 10 mg/g oral solution; AZD7594 1200 μg oral
Drug: AZD7594 Inhalation powder (400 μg) by DPI Device 1 (monodose inhaler) — Inhalation powder, hard capsules 400 μg Monodose inhaler; AZD7594 400 μg by dry powder inhaler (DPI) Device 1 (Monodose inhaler)
Drug: AZD7594 Inhalation powder (400 μg) by DPI device 2 (multiple-dose inhaler) — Inhalation powder, multiple-dose dry powder inhaler (DPI) 400 μg; AZD7594 400 μg by DPI Device 2 (multiple-dose DPI)
  Arms: Treatment sequence 1
Drug: AZD7594 Pressurized inhalation suspension (400 μg) by pMDI — Inhalation suspension 200 μg; AZD7594 400 μg by pressurized metered-dose inhaler (pMDI); 2 puffs x 200 μg = 400 μg
  Arms: Treatment sequence 2

SUMMARY:
This is an open-label,partially randomized, four-period study in healthy male subjects to assess the bioavailability and pharmacokinetics of a single dose of AZD7594 when administered intravenously, orally and inhaled via two different dry powder inhalers (DPIs) and a pressurized meter-dose inhaler (pMDI)

DETAILED DESCRIPTION:
This study is an open-label, partially randomized, 4-period, 5-treatment study in healthy male subjects, performed at a single study center. All subjects will receive the 4 of the 5 treatments. The IV infusion will be fixed as the first treatment (Period 1), the Monodose inhaler will be fixed as the second treatment (Period 2) and the oral formulation will be fixed as the fourth treatment (Period 4). During Period 3, subjects are split into 2 equal cohorts, multiple-dose DPI and pMDI.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male subjects aged 18 - 45 years with suitable veins for cannulation or repeated venipuncture.
3. Have a body mass index (BMI) between 18 and 30 kg/m2, inclusive, and weigh at least 50 kg.
4. Subjects should be willing to follow reproductive restrictions to prevent pregnancy and drug exposure of a female partner and refrain from donating sperm or fathering a child from the first day of dosing until 3 months after the last dose of investigational product.
5. Be able to inhale from the dry powder inhaler (DPI) devices and the pressurized metered-dose inhaler (pMDI) device according to given instructions.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, major medical/surgical procedure, or trauma within 4 weeks of the first administration of Investigational medicinal product (IMP).
4. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results at screening and check-in, as judged by the investigator.
5. Any clinically significant abnormal findings in vital signs after a 5 minute rest at screening and check-in, as judged by the investigator, defined as any of the following:

   * Systolic blood pressure (BP) > 140 mm Hg;
   * Systolic BP < 90 mm Hg;
   * Diastolic BP > 90 mm Hg;
   * Diastolic BP < 60 mm Hg; or
   * Heart rate < 40 or > 85 beats per minute (bpm).
6. Any clinically significant abnormities in physical examination or lung function, as judged by the investigator.
7. Any clinically significant abnormalities on 12-lead electrocardiogram (ECG) at screening and check-in, as judged by the investigator.
8. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc (QT interval corrected) interval changes. This includes subjects with any of the following:

   * Clinically significant PR (PQ) (ECG interval measured from the onset of the P wave to the onset of the QRS complex) interval prolongation;
   * Intermittent or persistent second or third degree AV block;
   * Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS (ECG interval measured from the onset of the QRS complex to the J point) > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of, for example, ventricular hypertrophy or pre-excitation; or
   * Abnormal T wave morphology, particularly in the protocol defined primary lead.
9. Prolonged QTcF (QT interval corrected for heart rate using Fridericia's formula) > 450 msec or family history of long QT (ECG interval measured from the onset of the QRS complex to the end of the T wave) syndrome.
10. Known or suspected history of drug abuse, as judged by the investigator
11. Current smokers or those who have smoked or used nicotine products within the previous 3 months.
12. History of alcohol abuse or excessive intake of alcohol as judged by the investigator.
13. Positive screen for drugs of abuse, alcohol, and cotinine at screening or on each admission to the study center.
14. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD7594 or to excipients.
15. Excessive intake of caffeine containing drinks e.g., coffee, tea, caffeine containing energy drinks and cola (in total no more than 3 cups per day).
16. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
17. Use of any prescribed or non-prescribed medication including vaccines, antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, vitamins and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life. Occasional use of paracetamol/acetaminophen is allowed for minor pains and headaches (no more than 3000 mg/day).
18. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
19. Has participated in a clinical study investigating clinical evaluation methods 1 month (or at least 5 half-lives) prior to the administration of investigational product.
20. Known Gilbert's syndrome, family history of Gilbert's syndrome or suspicion of Gilbert's syndrome based on liver function tests.
21. Any contraindication against the use of vagolytic or sympaticomimetic drugs, as judged by the investigator.
22. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
23. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) antibody.
24. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
25. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, M.D, Principal Investigator — Parexel
Locations (1):
- Research Site, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at PAREXEL International, Early Phase Clinical Unit, Baltimore, United States of America. A total of 30 subjects were enrolled in the study and Twenty-four subjects completed the study.
Pre-assignment Details: The IV infusion was fixed as the first treatment (Period 1), the monodose inhaler was fixed as the second treatment (Period 2) and the oral formulation was fixed as the fourth treatment (Period 4). During Period 3, subjects were split into 2 equal cohorts, multiple-dose DPI and pMDI.
Groups:
- IV, DPI 1, DPI 2, Oral: IV formulation, monodose inhaler, multiple-dose DPI, oral formulation
- IV, DPI 1, pMDI, Oral: IV formulation, monodose inhaler, pMDI, oral formulation
- pMDI (Additional): Pressurized metered-dose inhaler (pMDI)
Period: Overall Study
Arm/Group | IV, DPI 1, DPI 2, Oral | IV, DPI 1, pMDI, Oral | pMDI (Additional)
Started | 12 | 12 | 6
Completed | 9 | 9 | 6
Not Completed | 3 | 3 | 0
Not completed — Eligibility criteria not fulfilled | 0 | 2 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV, DPI 1, DPI 2, Oral | IV, DPI 1, pMDI, Oral | pMDI (Additional) | Total
Number analyzed (Participants) | 12 | 12 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.3 (7.07) | 31.3 (4.58) | 35.5 (2.88) | 32.9 (5.56)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 12 | 12 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) of AZD7594 Delivered by Monodose Inhaler and Multiple-dose DPI or pMDI in Terms of Pulmonary Bioavailability After Inhalation (Fpulmonary)
Description: For oral and inhalation administrations: pre-dose (0 hour) and post-dose at 15, 30 and 45 minutes and 1.0, 2.0, 4.0, 6.0, 8.0, 12.0, 16.0, 24.0, 36.0, 48.0, 72.0 and 96.0 hours following the administration of the investigational product AZD7594. For IV administration: pre-dose (0 hour) and post-dose at 5, 10, 15 (end of infusion), 30, 45, 60 and 90 minutes and 2.0, 4.0, 6.0, 8.0, 12.0, 16.0, 48.0, 72.0 and 96.0 hours following the start of the IV infusion of the investigational product AZD7594
Time Frame: 0-96 hours
Population: The PK analysis set will consist of all subjects in the safety analysis set for whom at least 1 PK parameters can be calculated for at least 1 treatment period and who have no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Groups:
- 400 µg DPI Device 1: AZD7594 400 μg delivered dose via Monodose inhaler
- 400 µg DPI Device 2: AZD7594 400 μg delivered dose via Multiple dose inhaler
- 400 µg pMDI: AZD7594 400 μg delivered dose pMDI
- 400 µg pMDI (Additional): AZD7594 400 μg delivered dose pMDI (Separate treatment)
Arm/Group | 400 µg DPI Device 1 | 400 µg DPI Device 2 | 400 µg pMDI | 400 µg pMDI (Additional)
Number analyzed (Participants) | 1 | 1 | 10 | 6
Percentage | 27.49 (NA) — Insufficient number of participants for CV%. | 30.73 (NA) — Insufficient number of participants for CV%. | NA (NA) — Plasma levels were too low to be detected hence not calculated. | NA (NA) — Plasma levels were too low to be detected hence not calculated.

2. Secondary Outcome: PK of AZD7594 Following Oral Administration by Assessment of the Absolute Systemic Bioavailability After Oral Administration (Fpo)
Description: as for outcome 1
Time Frame: 0-96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Groups:
- 150 µg IV Formulation: AZD7594 150 µg IV formulation
- 1200 µg Oral Formulation: AZD7594 1200 μg oral formulation
Arm/Group | 150 µg IV Formulation | 1200 µg Oral Formulation
Number analyzed (Participants) | 24 | 1
Percentage | NA (NA) — The Fpo is calculated only after oral administration hence not applicable for IV administration. | 0.4543 (NA) — The Fpo could not be calculated because the plasma levels after oral administration were so low, they could not be quantified.

3. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax)
Description: as for outcome 1
Time Frame: 0-96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | 400 µg DPI Device 1 | 400 µg DPI Device 2 | 400 µg pMDI | 400 µg pMDI (Additional) | 150 µg IV Formulation | 1200 µg Oral Formulation
Number analyzed (Participants) | 23 | 9 | 3 | 3 | 24 | 2
pmol/L | 112.6 (28.42) | 68.88 (22.16) | 13.93 (25.73) | 15.47 (11.34) | 6598 (27.05) | 19.31 (19.90)
Statistical Analysis 1: Comparison: 400 µg DPI Device 1 vs 400 µg DPI Device 2; Statistical Assessment of AZD7594 Pharmacokinetic Parameter (AUC0-t) Following Inhalation Administration ofAZD7594 via DPI Device 2 Versus DPI Device 1; Test type: Superiority or Other; Geometric mean ratio = 62.61, 90% CI 2-sided [53.01 to 73.94] — Ratio (%)

4. Secondary Outcome: Area Under the Plasma Concentration-curve From Time Zero to Time of Last Quantifiable Concentration (AUC0-t)
Description: as for outcome 1
Time Frame: 0-96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*pmol/L)
Arm/Group | 400 µg DPI Device 1 | 400 µg DPI Device 2 | 400 µg pMDI | 400 µg pMDI (Additional) | 150 µg IV Formulation | 1200 µg Oral Formulation
Number analyzed (Participants) | 23 | 9 | 1 | 3 | 24 | 1
(h*pmol/L) | 2524 (45.16) | 2648 (23.13) | 42.93 (NA) — Not applicable as n=1 | 572.7 (83.69) | 3343 (19.69) | 110.1 (NA) — Not applicable as n=1
Statistical Analysis 1: Comparison: 400 µg DPI Device 1 vs 400 µg DPI Device 2; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Geometric mean ratio = 101.15, 90% CI 2-sided [85.21 to 120.06] — Ratio (%)

5. Secondary Outcome: Absolute Systemic Bioavailability After Inhalation (F Inhalation, Total)
Description: as for outcome 1
Time Frame: 0-96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | 400 µg DPI Device 1 | 400 µg DPI Device 2 | 400 µg pMDI | 400 µg pMDI (Additional)
Number analyzed (Participants) | 23 | 9 | 1 | 6
Percentage | 28.21 (45.38) | 30.92 (20.87) | 0.3560 (NA) — Plasma levels were too low to be detected hence not calculated. | NA (NA) — Plasma levels were too low to be detected hence not calculated.

6. Secondary Outcome: Oral Bioavailability After Inhaled Treatment (F Oral)
Description: as for outcome 1
Time Frame: 0-96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | 400 µg DPI Device 1 | 400 µg DPI Device 2 | 400 µg pMDI | 400 µg pMDI (Additional)
Number analyzed (Participants) | 1 | 1 | 10 | 6
Percentage | 0.3294 (NA) — Not applicable as n=1 | 0.3147 (NA) — Not applicable as n=1 | NA (NA) — F oral was not calculated for the additional pMDI cohort as this cohort did not receive the oral and IV formulation treatments. | NA (NA) — F oral was not calculated for the additional pMDI cohort as this cohort did not receive the oral and IV formulation treatments.

7. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC)
Description: as for outcome 1
Time Frame: 0-96 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*pmol/L)
Arm/Group | 400 µg DPI Device 1 | 400 µg DPI Device 2 | 400 µg pMDI | 400 µg pMDI (Additional) | 150 µg IV Formulation | 1200 µg Oral Formulation
Number analyzed (Participants) | 23 | 9 | 10 | 6 | 24 | 9
(h*pmol/L) | NA (NA) — Not reported since parameter cannot be calculated as per standard criteria. | NA (NA) — Not reported since parameter cannot be calculated as per standard criteria. | NA (NA) — Plasma levels were too low to be detected hence not calculated. | NA (NA) — Plasma levels were too low to be detected hence not calculated. | 3465 (19.44) | NA (NA) — Plasma levels were too low to be detected hence not calculated.

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected from the signing of informed consent and AEs from check-in for the first treatment period until the final follow-up phone-call i.e., from Visit 1 to Visit 6 (Day -21 to Day 5).
Description: There were no deaths or SAEs reported in this study.
Groups:
- IV Formulation: AZD7594 150 μg IV formulation
- DPI Device 1: AZD7594 400 μg delivered dose monodose inhaler
- DPI Device 2: AZD7594 400 μg delivered dose multiple-dose DPI
- pMDI: AZD7594 400 μg delivered dose pMDI
- Oral Formulation: AZD7594 1200 μg oral formulation
- pMDI (Additional): AZD7594 400 μg delivered dose pMDI (separate treatment)
Arm/Group | IV Formulation | DPI Device 1 | DPI Device 2 | pMDI | Oral Formulation | pMDI (Additional)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/9 | 0/10 | 0/18 | 0/6
Other Adverse Events (participants affected / at risk) | 2/24 | 0/23 | 2/9 | 1/10 | 1/18 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Formulation (N=24) | DPI Device 1 (N=23) | DPI Device 2 (N=9) | pMDI (N=10) | Oral Formulation (N=18) | pMDI (Additional) (N=6)
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ocular hyperemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infusion site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Traumatic hematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.